CLINICAL TRIAL: NCT05462626
Title: Quality of Life and Occupational Performance in Community-Dwelling Older Adults: a Telehealth Lifestyle Pilot
Brief Title: A Telehealth Lifestyle Intervention for Community-Dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002841
Record Dates: First submitted 2022-06-28; First posted 2022-07-18 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-07

CONDITIONS: Lifestyle, Healthy; Quality of Life; Aging
Keywords: Occupational Therapy; Telehealth; Community Dwelling Older Adults; Health Literacy; Social Determinants of Health; Lifestyle Intervention

STUDY DESIGN:
Intervention Model Description: This quantitative pilot study will use a quasi-experimental approach with a single-group, pretest-posttest design to evaluate the effects of the Holistic Occupational Performance Empowerment (HOPE) lifestyle program on health-related quality of life and occupational performance of community-dwelling older adults.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- the Holistic Occupational Performance Empowerment (HOPE) Lifestyle Program (Experimental): The intervention will consist of six individualized sessions that will be conducted via a telehealth platform, each lasting about 45-60 minutes. Individual sessions allow for the participant's personal health factors to be discussed and reflected upon as the intervention is delivered weekly. Each week will comprise one or more lifestyle topics that are based on the twelve modules described in the Lifestyle Redesign® manual (Clark et al., 2015).
  Interventions: Behavioral: Holistic Occupational Performance Empowerment (HOPE) Lifestyle Program

INTERVENTIONS:
Behavioral: Holistic Occupational Performance Empowerment (HOPE) Lifestyle Program — The intervention is comprised of the following sessions and themes; Session 1: Informed Consent and Pre-Testing; Session 2: Occupation and Healthy Aging; Session 3: Longevity and Thriving; Session 4: Movement Matters; Session 5: Thoughtful Eating; Session 6: Stress and Sleep; Session 7: Navigating Health Care; Session 8: Post-Testing and Discharge.

SUMMARY:
The purpose of this study is to evaluate if an occupational therapy lifestyle program for community-dwelling older adults delivered individually through a telehealth platform can produce comparable outcomes in health-related qualify of life and occupational performance as found in studies that used a longer duration and group intervention.

DETAILED DESCRIPTION:
Eighty percent of older adult Americans live with at least one chronic disease and 70% manage two or more. Chronic diseases pose significant health and economic costs to individual older adults, burden families due to increased care dependency, and cause substantial strain on the healthcare system. Older adults residing in rural and non-urban communities in particular face additional health disparities due to lack of access or fewer options for health care services and providers. As one solution, telehealth can increase ease and access to health care services, deliver quality outcomes and comparable levels of satisfaction, and reduce costs for both the patient and the health care system. This quantitative pilot study will use a quasi-experimental approach with a single-group, pretest-posttest design to evaluate the effects of the Holistic Occupational Performance Empowerment (HOPE) lifestyle program to promote health-related quality of life and occupational performance of community-dwelling older adults.

Investigators anticipate recruiting 12 to 15 English-speaking, independent community-dwelling adults 65 years or older living in non-urban communities within 40 miles of Great Falls, Montana or Oregon City, Oregon. The participants will receive 1 goal-setting session in-person, 6 training sessions via telehealth, and 1 post-intervention debriefing session in-person across 8 weeks; each session will be 45-60 minutes. Each week will comprise one or more lifestyle topics that are based on the twelve modules described in the Lifestyle Redesign®️ manual. The sessions involve an introduction to a lifestyle topic with the investigator providing verbal and visual education, collaborative discussion and reflection, review of a participant's self-identified goals, recommendations and homework, and scheduling of the session for the subsequent week. By addressing health disparities and expanding access, occupational therapists will be more intentional in their delivery of telehealth lifestyle interventions and contribute to chronic disease prevention and reduction.

ELIGIBILITY:
Inclusion Criteria:

* Adults 65 years or older
* English-speaking
* Independent community-dwellers
* Living in non-urban communities within 40 miles of Great Falls, Montana or Oregon City, Oregon
* Self-reported adequate vision, with or without corrective lenses, to view and read paper-based and electronic materials with a minimum 12-point font size
* Demonstrate reasonable technology skills (e.g., access email and telehealth platform) with or without the help of a family member or caregiver
* Have consistent access to an electronic device that has Wi-Fi connection

Exclusion Criteria:

* Require any human assistance with activities of daily living
* Score of less than 12 out of 15 on 5-minute telephone version of the Montreal Cognitive Assessment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change Scores of 20-Item Short Form Survey | 2 Times; 1 Week Pre-Intervention; 1 Week Post-Intervention
  The 20-Item Short Form Survey (SF-20) is a shortened form of the original 36-item questionnaire created for the Medical Outcomes Study. The SF-20 utilizes close-ended, Likert-type questions to address self-reported health-related quality of life within six domains: physical functioning, role functioning, social functioning, mental health, current health perceptions, and pain. Raw scores from the 20 items are transformed linearly into 0-100 scales for each of the six domains. Higher scores indicate better physical, role, and social functioning, better mental health and health perceptions, and more pain.
Change Scores of Goal Attainment Scaling | 2 Times; 1 Week Pre-Intervention; 1 Week Post-Intervention
  Goal attainment scaling (GAS) is a method of scoring the extent to which a participant's individualized goals are achieved over the course of an intervention. The participants will be asked to identify three occupation-based, lifestyle-focused SMART (specific, measurable, attainable, realistic, and timely) goals. Goals are weighted based on the participant's rating of importance and level of difficulty on a scale of 0 to 3 where higher scores indicate greater importance and greater difficulty, respectively. Each goal is also rated on a 5-point scale capturing a degree of attainment, the expected outcome at pre-intervention, and the achieved outcome at post-intervention. Scores can range from -2 to +2 where a median score of 0 indicates goals were achieved as expected, negative scores indicate goals with worse than expected outcomes, and positive scores indicate goals with better than expected outcomes.
The Short Assessment of Health Literacy-English (SAHL-E) | 1 Week Pre-Intervention
  The Short Assessment of Health Literacy-English (SAHL-E) is an 18-item test designed to help health professionals assess the ability of English-speaking adults to read and understand common medical terms. Participants score between 0 and 18 points with higher scores indicating better health literacy. Scores of 14 or below indicate low health literacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amdie, F. Z., & Woo, K. (2020). The use of mHealth technology for chronic disease management: The challenges and opportunities for practical application. Wounds International, 11(2), 32-38. https://www.woundsinternational.com/resources/details/the-use-of-mhealth-technology-for-chronic-disease-management-the-challenges-and-opportunities-for-practical-application
- [Background] Arain M, Campbell MJ, Cooper CL, Lancaster GA. What is a pilot or feasibility study? A review of current practice and editorial policy. BMC Med Res Methodol. 2010 Jul 16;10:67. doi: 10.1186/1471-2288-10-67. PMID 20637084
- [Background] Cahill, S. (2021). Research update on telehealth: Client outcomes and satisfaction, occupation-based coaching, and stroke rehabilitation. American Occupational Therapy Association. https://www.aota.org/publications/ot-practice/ot-practice- issues/2021/research-update-telehealth
- [Background] Centers for Disease Control and Prevention. (2009). The power of prevention: Chronic disease...the public health challenge of the 21st century. National Center for Chronic Disease Prevention and Health Promotion. https://www.cdc.gov/chronicdisease/pdf/2009-power-of-prevention.pdf
- [Background] Clark F, Azen SP, Zemke R, Jackson J, Carlson M, Mandel D, Hay J, Josephson K, Cherry B, Hessel C, Palmer J, Lipson L. Occupational therapy for independent-living older adults. A randomized controlled trial. JAMA. 1997 Oct 22-29;278(16):1321-6. PMID 9343462
- [Background] Clark, F. A., Blanchard, J., Sleight, A., Cogan, A., Florindez, L., Gleason, S., Heymann, R., Hill, V., Holden, A., Murphy, M. Proffitt, R., Schepens Niemiec, S., & Vigen, C. (2015). Lifestyle Redesign: The intervention tested in the USC Well Elderly Studies (2nd ed.) Bethesda, MD: AOTA Press.
- [Background] Clark F, Jackson J, Carlson M, Chou CP, Cherry BJ, Jordan-Marsh M, Knight BG, Mandel D, Blanchard J, Granger DA, Wilcox RR, Lai MY, White B, Hay J, Lam C, Marterella A, Azen SP. Effectiveness of a lifestyle intervention in promoting the well-being of independently living older people: results of the Well Elderly 2 Randomised Controlled Trial. J Epidemiol Community Health. 2012 Sep;66(9):782-90. doi: 10.1136/jech.2009.099754. Epub 2011 Jun 2. PMID 21636614
- [Background] Edmonds, W. A., & Kennedy, T. D. (2010). A reference guide to basic research design: A visual system for research design in education and the social and behavioral sciences. Pearson Learning Solutions.
- [Background] Gately ME, Trudeau SA, Moo LR. Feasibility of Telehealth-Delivered Home Safety Evaluations for Caregivers of Clients With Dementia. OTJR (Thorofare N J). 2020 Jan;40(1):42-49. doi: 10.1177/1539449219859935. Epub 2019 Jul 18. PMID 31319745
- [Background] Lee SY, Stucky BD, Lee JY, Rozier RG, Bender DE. Short Assessment of Health Literacy-Spanish and English: a comparable test of health literacy for Spanish and English speakers. Health Serv Res. 2010 Aug;45(4):1105-20. doi: 10.1111/j.1475-6773.2010.01119.x. Epub 2010 May 24. PMID 20500222
- [Background] National Council on Aging. (2021). Get the facts on healthy aging. https://www.ncoa.org/article/get-the-facts-on-healthy-aging
- [Background] Nesreddine, Z. (2021). Mini Montreal Cognitive Assessment (Mini MoCA) version 2.1: Administration and scoring instructions. www.mocatest.org
- [Background] Portney, L. G. (2020). Foundations of clinical research (4th ed.). FA Davis.
- [Background] RAND Corporation. (n.d.). More about the 20-item short form survey (SF-20). https://www.rand.org/health-care/surveys_tools/mos/20-item-short-form/more.html
- [Background] Rural Health Information Hub. (2019). Rural health disparities. Health Resources and Services Administration, United States Department of Health and Human Services https://www.ruralhealthinfo.org/topics/rural-health-disparities#causes
- [Background] Solomon GM, Bailey J, Lawlor J, Scalia P, Sawicki GS, Dowd C, Sabadosa KA, Van Citters A. Patient and family experience of telehealth care delivery as part of the CF chronic care model early in the COVID-19 pandemic. J Cyst Fibros. 2021 Dec;20 Suppl 3:41-46. doi: 10.1016/j.jcf.2021.09.005. PMID 34930542
- [Background] Stolee P, Zaza C, Pedlar A, Myers AM. Clinical experience with Goal Attainment Scaling in geriatric care. J Aging Health. 1999 Feb;11(1):96-124. doi: 10.1177/089826439901100106. PMID 10848144
- [Background] Tenforde AS, Borgstrom H, Polich G, Steere H, Davis IS, Cotton K, O'Donnell M, Silver JK. Outpatient Physical, Occupational, and Speech Therapy Synchronous Telemedicine: A Survey Study of Patient Satisfaction with Virtual Visits During the COVID-19 Pandemic. Am J Phys Med Rehabil. 2020 Nov;99(11):977-981. doi: 10.1097/PHM.0000000000001571. PMID 32804713
- [Background] Turner-Stokes L. Goal attainment scaling (GAS) in rehabilitation: a practical guide. Clin Rehabil. 2009 Apr;23(4):362-70. doi: 10.1177/0269215508101742. Epub 2009 Jan 29. PMID 19179355